CLINICAL TRIAL: NCT02930473
Title: Short-term Efficacy Evaluation of a Psychotherapeutic Intervention Model in Nursing on Nursing Diagnosis "Anxiety": A Randomised Controlled Trial
Brief Title: Evaluation of a Psychotherapeutic Intervention Model in Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Miguel Correia Sampaio (Other)
Responsible Party: Sponsor-Investigator, Francisco Miguel Correia Sampaio, RMN, MSc, PhD Student, Universidade do Porto
Organization: Universidade do Porto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICBAS 1988
Record Dates: First submitted 2016-02-05; First posted 2016-10-12 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Anxiety
Keywords: Psychotherapy; Nursing; Nursing Care; Nursing Model; Randomised Controlled Trial
MeSH Terms: conditions — Anxiety Disorders | interventions — Psychotropic Drugs

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychotherapeutic Intervention(s) for Anxiety (Experimental): People diagnosed with "Anxiety" (according to ICNP/NANDA standardized nursing language) will be treated using Nursing Interventions Classification (NIC) psychotherapeutic intervention(s) for anxiety (plus psychopharmaceuticals).
  Interventions: Behavioral: NIC Psychotherapeutic Intervention(s) for Anxiety; Drug: Psychopharmaceuticals (any drugs prescribed by the psychiatrist)
- Treatment-as-Usual for Anxiety (Active Comparator): People diagnosed with "Anxiety" (according to ICNP/NANDA standardized nursing language) will receive treatment as usual for anxiety (psychopharmaceuticals).
  Interventions: Drug: Psychopharmaceuticals (any drugs prescribed by the psychiatrist)

INTERVENTIONS:
Behavioral: NIC Psychotherapeutic Intervention(s) for Anxiety — Patients will be treated by NIC psychotherapeutic intervention(s) for anxiety (e.g. anxiety reduction) plus psychopharmaceuticals prescribed by their psychiatrist.
  Arms: Psychotherapeutic Intervention(s) for Anxiety
Drug: Psychopharmaceuticals (any drugs prescribed by the psychiatrist) — Patients will be treated only by psychopharmaceuticals prescribed by their psychiatrist.

SUMMARY:
This study aims to evaluate the efficacy of a psychotherapeutic intervention model in nursing on the nursing diagnosis "Anxiety". A randomised controlled trial will be carried out to do so.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of a psychotherapeutic intervention model in nursing on nursing diagnosis "Anxiety" (according to International Classification for Nursing Practice (ICNP)/North American Nursing Diagnoses Association (NANDA) standardized nursing language). A randomised controlled trial will be carried out to do so. In a single-blinded nurse-led 6 months controlled trial, conducted at a hospital outpatient setting in Portugal, approximately 60 patients with anxiety will be randomised to the intervention (n=30) or control groups (n=30). The objective is to compare the outcomes associated with "treatment-as-usual" and the benefits of implementing the psychotherapeutic intervention model in nursing previously developed (5 sessions), which will be evaluated using Nursing Outcomes Classification (NOC) outcomes "Anxiety Level" and "Anxiety Self-Control" (Portuguese version).

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old;
* Nursing Diagnosis "Anxiety" (according to ICNP/NANDA standardized nursing language) - assessment using NOC outcome "Anxiety Level" (Portuguese version);
* Elementary education (completed).

Exclusion Criteria:

* Psychiatric diagnosis of dementia or psychotic spectrum disorder;
* Being in therapy provided by a psychologist (at the moment of the session 0);
* Cognitive impairment (assessment using Mini-Mental State Examination);
* Moderate or severe intellectual disability;
* Confusional state;
* Psychomotor agitation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in the Level of Anxiety (NOC outcomes "Anxiety Level" and "Anxiety Self-Control" - Portuguese version) | At the beginning of the study (Session 0) and one week after session 5 (approximately 6 weeks after the beginning of the study)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Sampaio, MSc, Principal Investigator — Instituto de Ciências Biomédicas Abel Salazar da Universidade do Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sampaio FMC, Araujo O, Sequeira C, Lluch Canut MT, Martins T. A randomized controlled trial of a nursing psychotherapeutic intervention for anxiety in adult psychiatric outpatients. J Adv Nurs. 2018 May;74(5):1114-1126. doi: 10.1111/jan.13520. Epub 2018 Jan 25. PMID 29288510